CLINICAL TRIAL: NCT07190911
Title: Efficacy of Olfactive Training on Loss of Smell and Taste Caused by SARS CoV2 (Covid-Smell)
Brief Title: Efficacy of Olfactive Training on Loss of Smell and Taste Caused by SARS CoV2 COVID-19 (Covid-Smell)
Acronym: COVID-SMELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PAP_RI2_2020/17; 2020-A02606-33 (Registry Identifier: ANSM)
Record Dates: First submitted 2025-09-22; First posted 2025-09-24 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: COVID - 19
Keywords: Covid-19; olfactory training; olfactory and taste loss
MeSH Terms: conditions — COVID-19; Anosmia; Ageusia

STUDY DESIGN:
Intervention Model Description: To prove this efficiency, a parallel prospective comparative study appear to be one of the best the way.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- olfactory training arm (Experimental): with a daily olfactory training during 2 month
  Interventions: Other: Olfactory rehabilitation consists of smelling a series of spices every day for 2 months
- no olfactory training (No Intervention)

INTERVENTIONS:
Other: Olfactory rehabilitation consists of smelling a series of spices every day for 2 months — Olfactory rehabilitation consists of smelling a series of spices every day for 2 months: vanilla, coffee, dill, thyme, cinnamon, cloves, lavender, coriander, light vinegar, mint, and cumin.
  This rehabilitation is based on the protocols proposed by SFORL (French ORL society) and Oleszkiewicz et al.8
  Allergies to certain spices will be noted at the start of the study:
  * in known allergy: change by another spice which belongs to the same chemical category.
  * in case of allergies to several scents: patient is not included in the study.
  * in case of allergy appearing during participation: clinical evaluation by ENT, change by another spice which belongs to the same chemical category.
  * in case of allergies to several scents occuring during participation: patient is excluded from the study.
  Arms: olfactory training arm

SUMMARY:
The purpose of this study is to evaluate efficiency of two months of olfactive training on olfactory and taste loss secondary to covid-19. We will compare 2 groups : olfactive training group versus no olfactive training group.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate efficiency of two months of olfactive training on olfactory and taste loss secondary to covid-19. We will compare 2 groups : olfactive training group versus no olfactive training group.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 infection suspect or confirmed
* supported by CHU Guadeloupe
* with brutal olfactory or taste loss
* affiliated or beneficiary of a social security scheme
* informed consent signed

Exclusion Criteria:

* recent rhinosinusitis, less than 6 months
* lingual pathology
* communication disorder
* Patients subject to a justice safeguard
* Allergy to several spices that are part of the rehabilitation set
* Pregnant or breastfeeding women
* Absence of signed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2022-03-09 (Actual)

PRIMARY OUTCOMES:
Taste and Smell Survey (TSS). | Baseline and 2 months
  Patients will have this auto evaluation scale at the inclusion (D0) and 2 month after inclusion (D60).

SECONDARY OUTCOMES:
Sniffin' stick test : | 2 month
  The Sniffin' Stick Test assesses the sense of smell by measuring odor detection threshold, discrimination, and identification, and is used for diagnosing and monitoring olfactory disorders.
Olfaction and taste evolution evaluated with a daily visual scale | Every day from inclusion to 2 months
  Visual analogue scale from 0 to 10 to assess dysosmia and dysgeusia, with 0 indicating normal function and 10 indicating complete deficit.

CONTACTS AND LOCATIONS:
Overall Officials: Suzy Duflo, MD PhD, Principal Investigator — CHU de la Guadeloupe
Locations (1):
- Chu de La Guadeloupe, Pointe-à-Pitre, Guadeloupe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Medical thesis of Ms. Nordera, entitled "Study on the Effectiveness of Olfactory Rehabilitation for Dysosmia and Dysgeusia Following SARS-CoV-2 Infection — https://dumas.ccsd.cnrs.fr/dumas-04551904